CLINICAL TRIAL: NCT06455631
Title: The Effect of Facilitated Tucking, Oral Breast Milk, and Kangaroo Care on Pain During Band Removal in Preterm Newborns
Brief Title: The Effect of Non-pharmacological Methods on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Negarin Akbari, Assisstant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-10840098-202.3.02-3029
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pain; Infant ALL; Preterm
Keywords: Preterm Infant; Oral Breast Milk; Fetal Position; Kangaroo Care; Band Removal; Pain
MeSH Terms: conditions — Pain; Premature Birth | interventions — Facilitated Tucking; Milk, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Breast Milk and Facilitated Tucking (Experimental): In the facilitated tucking position + oral breast milk group, preterm newborns will be placed in the facilitated tucking position by the researcher 15 minutes before the tape removal procedure and given oral breast milk 2 minutes before the tape removal procedure. The facilitated tucking position will be maintained until 2 minutes after the tape removal procedure. To prevent heat loss, the preterm newborns will be placed in the fetal position inside the incubator by using the incubator windows without opening the incubator lid.
  Interventions: Procedure: Facilitated Tucking, Oral Breast Milk , Kangaroo Care
- Kangaroo Care and Oral Breast Milk Odor (Experimental): In the kangaroo care + oral breast milk group, preterm newborns will undergo kangaroo care 15 minutes prior to tape removal and receive oral breast milk 2 minutes before. During kangaroo care, mothers can interact with their babies but cannot feed them. After ensuring comfort, this position will be maintained for 15 minutes before tape removal. The nurse will then remove the tape while the baby is in kangaroo care, followed by an additional 2 minutes of kangaroo care. Kangaroo care can continue post-data collection based on maternal preference, baby's condition, and clinical circumstances.
  Interventions: Procedure: Facilitated Tucking, Oral Breast Milk , Kangaroo Care
- Control (No Intervention): The newborns in the control group will undergo the routine nesting procedure of the clinic. All newborns will be placed in the lateral position. For ethical reasons, if babies cry during or after the procedure, gentle touch and verbal comfort will be provided to them.

INTERVENTIONS:
Procedure: Facilitated Tucking, Oral Breast Milk , Kangaroo Care — Before data collection, the researcher will inform families of newborns meeting the sample criteria about the study and obtain written consent from participating parents. Newborn and parent information will be recorded. Procedures will occur between 08:00 and 16:00, with one researcher, two nurses, and a preterm newborn present during tape removal. Tape removal will be done by the same nurse. Physiological and behavioral responses will be recorded before, during, and after tape removal. Breast milk will be orally administered during tape removal, with the amount adjusted based on gestational age. Measurements will be taken at specified time points, including heart rate, respiratory rate, oxygen saturation, and PIPP-R score. These procedures will also apply to the control group. PIPP-R scores will be recorded by two evaluators based on video recordings.
  Arms: Kangaroo Care and Oral Breast Milk Odor; Oral Breast Milk and Facilitated Tucking

SUMMARY:
The research will be conducted using a randomized controlled experimental method.The preterm newborns included in the study will be randomized into three groups using the sealed envelope method. In the facilitated tucking position + oral breast milk group, preterm newborns will be placed in the facilitated tucking position 15 minutes before tape removal and given oral breast milk 2 minutes before. This position will be maintained until 2 minutes after tape removal. Preterm newborns in the kangaroo care + oral breast milk group will undergo kangaroo care 15 minutes before tape removal and receive oral breast milk 2 minutes before. Kangaroo care allows mother-baby interaction but no feeding. In the control group, newborns will undergo routine nesting with gentle touch and verbal comfort provided if they cry.This study is designed to evaluate the effect of the fetal position, oral breast milk administration, and kangaroo care on pain during tape removal in preterm newborns.

DETAILED DESCRIPTION:
In the study, the groups of the babies will be determined by a lottery method. Preterm babies included in the study will be randomly assigned to three groups using a closed envelope method. To ensure equal distribution of babies according to gestational age, two sets of envelopes will be created for 30-33+6 weeks and 34-36+6 weeks. An independent nurse working in the NICU will be asked to select a paper from the closed envelope corresponding to the baby's gestational week. Based on the number written on the selected paper, the baby will be included in the study group. The groups will be: Group 1 - facilitated tucking position + oral breast milk, Group 2 - kangaroo care + oral breast milk, and Group 3 - control group. After the babies are assigned to the groups, data collection will begin.

Before data collection, the researcher will provide necessary information about the study to the families of the newborns who meet the sample selection criteria and will answer their questions. After obtaining written consent from the parents of the babies who agree to participate, they will be included in the study. The information in the introductory information form for the newborn and parents will be recorded by the researcher.

1. Breast Milk Administration Procedure During tape removal, babies will be given breast milk orally. The amount of milk given to the baby will be adjusted according to gestational age (1.5 ml for 30+1-32 weeks; 2 ml for 32+1-36+6 weeks) (Peng et al., 2018).
2. Tape Removal Procedure The same product (medical tape suitable for the baby and causing minimal tissue trauma) will be used to effectively secure medical devices. To remove the tape, moistened gauze or saline pads will be used to gently and slowly remove it parallel to the skin surface horizontally.

1. GROUP: Interventions for the Facilitated Tucking Position + Oral Breast Milk Group Preterm newborns in the facilitated tucking position + oral breast milk group will be placed in the facilitated tucking position by the researcher 15 minutes before the tape removal procedure and given oral breast milk 2 minutes before the tape removal procedure. The facilitated tucking position will be maintained until 2 minutes after the tape removal procedure. To prevent heat loss, preterm newborns will be positioned in the right lateral position inside the incubator by using the incubator windows without opening the incubator lid, with their arms and legs brought to the midline in the facilitated tucking position.

2. GROUP: Interventions for the Kangaroo Care + Oral Breast Milk Group Preterm newborns in the kangaroo care + oral breast milk group will receive kangaroo care from the researcher 15 minutes before the tape removal procedure to alleviate pain; oral breast milk will be given 2 minutes before the tape removal procedure. The mothers of the babies in this group will be seated in the neonatal intensive care unit (NICU), and a nurse will place the newborn upright between the mother's bare breasts, slightly extending the head to facilitate breathing. The legs will be spread under the mother's chest and positioned in flexion. The back will be wrapped with extra fabric up to the ear level to prevent heat loss. During the contact, the mother will be allowed to talk to, move, or engage in other activities with her baby, but feeding will not be permitted. After ensuring the comfort of both the newborn and the mother, this position will be maintained for 15 minutes before the tape removal procedure. Subsequently, the nurse will perform the tape removal while the newborn is in the kangaroo care position, and the mother and baby will remain in kangaroo care for an additional 2 minutes. Once data collection is complete, kangaroo care can continue based on the mother's wishes, the baby's condition, and clinical circumstances.

Interventions for the CONTROL Group Newborns in the control group will undergo the routine nesting procedure of the clinic. All newborns will be placed in the lateral position. For ethical reasons, if babies cry during or after the procedure, gentle touch and verbal comfort will be provided to them.

In all experimental groups, heart rate, respiratory rate, oxygen saturation values, and PIPP-R scores will be measured and recorded at the following time points:

* 0 minutes: Measurements will be taken and recorded immediately before any intervention while the baby is in a resting position. Then, depending on the baby's group, either the facilitated tucking position or kangaroo care will be applied.
* 13 minutes: Measurements will be taken and recorded immediately before giving oral breast milk.
* 15 minutes: Measurements will be taken and recorded during the tape removal procedure.
* 17 minutes: Measurements will be taken and recorded 2 minutes after the tape removal procedure, while non-pharmacological interventions continue.
* In the control group, similar measurements and assessments will be conducted at the same time intervals and recorded.

The PIPP-R scores of all groups will be recorded on a data assessment form by two independent evaluators based on video recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between 30 and 36+6 weeks
2. The newborn not having undergone a painful procedure at least 1 hour before the intervention
3. Not having received analgesic and/or sedative medication in the last hour
4. Presence of maternal breast milk
5. Not having received oral or enteral feeding in the last hour
6. Not receiving continuous positive airway pressure (CPAP) or oxygen therapy

Exclusion Criteria:

1. Having ventilator support
2. Having a congenital anomaly
3. Undergoing continuous sedative treatment
4. Having a congenital malformation that could cause asphyxia and affect breathing
5. Having intracranial hemorrhage

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Pain in preterm infant | Maximum 17 minutes
  We will assess newborns' pain using the PIPP-R tool before the procedure and at 13, 15, and 17 minutes after starting the procedure.

SECONDARY OUTCOMES:
Heart rate | Maximum 17 minutes
  In order to determine the infant's heart rate, a 'Covidien' pulse oximeter will be used. It will be recorded by the observing nurse in the observation form before the procedure and at 13, 15, and 17 minutes after starting the procedure.
Oxygen Saturation | Maximum 17 minutes
  In order to determine the infant's oxygen saturation, a 'Covidien' pulse oximeter will be used. It will be recorded by the observing nurse in the observation form before the procedure and at 13, 15, and 17 minutes after starting the procedure.
Respiratory rate | Maximum 17 minutes
  A Casio brand stopwatch will be used to count the respiratory rate of the preterm newborn.

CONTACTS AND LOCATIONS:
Overall Officials: Cana Genç, Ph.D student, Principal Investigator — Fenerbahce University; Duygu Gözen, Ph.D, Study Chair — Koç University; İrem Baylı, Ms.C, Principal Investigator — Medipol hospital; Ayhan Taştekin, Dr, Principal Investigator — Medipol hospital; Negarin Akbari, Study Chair — Department of Nursing, Faculty of Health Sciences, Fenerbahce University, Istanbul, Turkey
Locations (1):
- Fenerbahce University, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No